CLINICAL TRIAL: NCT04629950
Title: A Pilot Study of Rimegepant in Moderate Plaque-type Psoriasis
Brief Title: Rimegepant in Moderate Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-07022368
Record Dates: First submitted 2020-11-11; First posted 2020-11-16 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Rimegepant (Experimental): Participants receive a rimegepant 75 mg tablet orally every other day for 16 weeks.
  Interventions: Drug: Rimegepant
- Placebo (Placebo Comparator): Participants receive a placebo tablet matching rimegepant orally every other day for 16 weeks.
  Interventions: Drug: Placebo
- Rimegepant Extension-Previously Received Rimegepant-Open Label (Experimental): Participants who previously received rimegepant receive a rimegepant 75 mg tablet orally every other day for an additional 12 weeks.
  Rimegepant: Active Agent
  Interventions: Drug: Rimegepant
- Rimegepant Extension-Previously Received Placebo-Open Label (Experimental): Participants who previously received placebo receive a rimegepant 75 mg tablet orally every other day for an additional 12 weeks.
  Rimegepant: Active Agent
  Interventions: Drug: Rimegepant

INTERVENTIONS:
Drug: Rimegepant — Active Agent
  Other Names: Nurtec
  Arms: Rimegepant; Rimegepant Extension-Previously Received Placebo-Open Label; Rimegepant Extension-Previously Received Rimegepant-Open Label
Drug: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the use of a new investigational medication for the treatment of moderate plaque-type psoriasis. The study medication is rimegepant, an orally administered small molecule competitive inhibitor of the calcitonin gene-related peptide (CGRP) receptor. This medication, rimegepant, has been approved by the FDA under the trade name Nurtec for the treatment of acute migraine. However, rimegepant has not been studied in the treatment of moderate plaque-type psoriasis and is investigational for this indication.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study of rimegepant 75 mg dosed every other day for the treatment of mild to moderate psoriasis. Subjects must have at 3% body surface area involvement before entry into the study. Psoriasis Area and Severity Index (PASI) and Investigator's Global Assessment (IGA) scores will be calculated and subjects will each complete the Dermatology Life Quality Index (DLQI) instrument as well an itch assessments. These assessments will be performed at baseline and every 2 weeks in follow-up. Areas of psoriasis in each subject will be photographed at baseline and two very similar appearing lesions identified for biopsy of one on day 1 and the other at the end of week 16. Patients will also repeat the DLQI at each visit. Subjects will also be photographed at each visit. Subjects will discontinue medications after the end of week 16. Subjects who complete the 20-week protocol will have the option of entering a 3-month, open-label extension of the study in which they will take 75 mg of rimegepant every other day for an additional 12 weeks. Eligible subjects have 2 weeks past visit 11 to enroll in the extension. For those rolling over before visit 11, visits 11 and 12 can be combined. They will have the same 7 assessments as in the previous portion of the study every 4 Protocol #20-07022368 Version Date 5/10/24 weeks including an EKG. The inclusion and exclusion criteria remain the same.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with at least 3% body surface are involved with psoriasis and a PASI score >5.
* Between 18 and 75 years of age.
* Documentation of a definite diagnosis of psoriasis by a dermatologist or biopsy.
* For women of childbearing potential, a negative urine pregnancy test within 48 hours of randomization. Female subjects should not have attempted to become pregnant in the month prior to exposure to rimegepant and agree not to attempt to become pregnant for 8 weeks after exposure to rimegepant.
* A valid form of contraception must be documented for men and women of child-bearing potential.

  * The two methods for women of childbearing potential should include:

    * One barrier method (for example, Diaphragm with spermicidal gel, condom with spermicidal gel, cervical caps or intrauterine devices placed for at least four weeks before sexual intercourse); AND
    * One additional method. The other method could include hormonal contraceptives, or second barrier method as listed above.
  * The two options for men of childbearing potential should include:

    * Simultaneous use of male condom, and for the female partner, hormonal contraceptives (for example, birth control pills, implants, patch, depot injection, used since at least 4 weeks) or intra-uterine contraceptive device (placed since at least 4 weeks) before sexual intercourse; OR simultaneous use of male condom, and for the female partner, diaphragm with intravaginally applied spermicide.

Exclusion Criteria:

* Any ongoing medical illness or condition that places the participant at higher risk for adverse outcomes or inability to complete study procedures in the opinion of the study investigator.
* Pregnancy or breastfeeding.
* Known autoimmune disorders other than psoriasis.
* Current use of corticosteroids or immunosuppressive medications (for any reason).
* Immunodeficiency diseases.
* Use of any biologic agent/monoclonal antibody within 5 half-lifes prior to baseline.
* Ultraviolet light treatment, cyclosporine, oral corticosteroids, methotrexate, oral retinoids, mycophenolate mofetil, thioguanine, hydroxyurea, sirolimus or azathioprine within the 4 weeks prior to baseline or had topical psoriasis treatment within the previous 2 weeks prior to baseline.
* Participation in another clinical trial involving an investigational drug within the last 30 days prior to baseline.
* Inability for woman of child-bearing potential to use an effective form of contraception if sexually active.
* Use of any medication that is a strong or moderate inhibitor of CYP3A, a strong or moderate inducer of CYP3A, or an inhibitor of glycoprotein (P-gp) or Breast Cancer Resistance Protein (BCRP). Please see Section 7.8 for more information.
* Subject history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Subjects with myocardial infarction (MI), acute coronary syndrome (ACS), percutaneous coronary intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during 6 months (24 weeks) prior to screening.
* Uncontrolled hypertension or uncontrolled diabetes (however, subjects can be included who have stable hypertension and/or diabetes for 3 months (12 weeks) prior to screening). Blood pressure greater than 150 mm Hg systolic or 100 mm Hg diastolic after 10 minutes of rest is exclusionary
* Subjects with an active episode of major depressive episode within the last 6 months are ineligible. Subjects with major depressive disorder or any anxiety disorder are eligible only if they are on stable medication for each disorder for at least 3 months prior to the Screening visit.
* Subject has a history or diagnosis of Gilbert's Syndrome or any other active hepatic or biliary disorder
* Hematologic or solid malignancy diagnosis within 5 years prior to screening. Subjects with a history of localized basal cell or squamous cell skin cancer are eligible for the study if they are cancer-free prior to the screening visit in this study.
* Subject has current diagnosis of major depressive disorder requiring treatment with atypical antipsychotics, schizophrenia, bipolar disorder, or borderline personality disorder.
* History of gallstones.
* Subject has current diagnosis of major depressive disorder requiring treatment with atypical antipsychotics, schizophrenia, bipolar disorder, or borderline personality disorder.
* The use of CGRP antagonists (biologic [e.g. Aimovig™, Emgality® and Ajovy™, VyeptiTM] or small molecule [ e.g. Ubrelvy™ {ubrogepant]]) other than rimegepant is prohibited during the study.
* Concomitant use of atypical antipsychotics such as Abilify (aripiprazole), Zyprexa (olanzapine), Seroquel (quetiapine), Geodon (ziprasidone), or Risperdal (risperidone).
* Depakote/Depakene (divalproex/valproic acid/valproate) is prohibited during the study.
* Concomitant use of LAMICTAL (lamotrigine) is prohibited during the study.
* Concomitant use of Modafinil (PROVIGIL®) is prohibited during the study.
* Exclusionary screening lab test findings:

  * Serum bilirubin (Total, Direct or Indirect) > 1 x ULN (Only abnormal values of between 1-1.5x ULN may be repeated once for assessment of eligibility prior to randomization)
  * AST or ALT > 1 x ULN (Only abnormal values of between 1-1.5x ULN may be repeated once for assessment of eligibility prior to randomization)
  * Neutrophil count ≤ 1000/μL (or equivalent)
  * HbA1c > 6.5%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Granstein, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Weill Cornell Medicine, New York, New York
  - Sadick Dermatology, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajguru JP, Maya D, Kumar D, Suri P, Bhardwaj S, Patel ND. Update on psoriasis: A review. J Family Med Prim Care. 2020 Jan 28;9(1):20-24. doi: 10.4103/jfmpc.jfmpc_689_19. eCollection 2020 Jan. PMID 32110559
- [Background] Takeshita J, Grewal S, Langan SM, Mehta NN, Ogdie A, Van Voorhees AS, Gelfand JM. Psoriasis and comorbid diseases: Implications for management. J Am Acad Dermatol. 2017 Mar;76(3):393-403. doi: 10.1016/j.jaad.2016.07.065. PMID 28212760
- [Background] Greb JE, Goldminz AM, Elder JT, Lebwohl MG, Gladman DD, Wu JJ, Mehta NN, Finlay AY, Gottlieb AB. Psoriasis. Nat Rev Dis Primers. 2016 Nov 24;2:16082. doi: 10.1038/nrdp.2016.82. PMID 27883001
- [Background] Kaushik SB, Lebwohl MG. Review of safety and efficacy of approved systemic psoriasis therapies. Int J Dermatol. 2019 Jun;58(6):649-658. doi: 10.1111/ijd.14246. Epub 2018 Sep 23. PMID 30246393
- [Background] Racz E, Prens EP. Phototherapy of Psoriasis, a Chronic Inflammatory Skin Disease. Adv Exp Med Biol. 2017;996:287-294. doi: 10.1007/978-3-319-56017-5_24. PMID 29124709
- [Background] Farber EM, Lanigan SW, Boer J. The role of cutaneous sensory nerves in the maintenance of psoriasis. Int J Dermatol. 1990 Jul-Aug;29(6):418-20. doi: 10.1111/j.1365-4362.1990.tb03825.x. PMID 2397964
- [Background] Zhu TH, Nakamura M, Farahnik B, Abrouk M, Lee K, Singh R, Gevorgyan A, Koo J, Bhutani T. The Role of the Nervous System in the Pathophysiology of Psoriasis: A Review of Cases of Psoriasis Remission or Improvement Following Denervation Injury. Am J Clin Dermatol. 2016 Jun;17(3):257-63. doi: 10.1007/s40257-016-0183-7. PMID 26935938
- [Background] Perlman HH. Remission of psoriasis vulgaris from the use of nerve-blocking agents. Arch Dermatol. 1972 Jan;105(1):128-9. doi: 10.1001/archderm.1972.01620040088028. No abstract available. PMID 5009614
- [Background] Aschenbeck KA, Hordinsky MK, Kennedy WR, Wendelschafer-Crabb G, Ericson ME, Kavand S, Bertin A, Dykstra DD, Panoutsopoulou IG. Neuromodulatory treatment of recalcitrant plaque psoriasis with onabotulinumtoxinA. J Am Acad Dermatol. 2018 Dec;79(6):1156-1159. doi: 10.1016/j.jaad.2018.07.058. No abstract available. PMID 30420008
- [Background] Ostrowski SM, Belkadi A, Loyd CM, Diaconu D, Ward NL. Cutaneous denervation of psoriasiform mouse skin improves acanthosis and inflammation in a sensory neuropeptide-dependent manner. J Invest Dermatol. 2011 Jul;131(7):1530-8. doi: 10.1038/jid.2011.60. Epub 2011 Apr 7. PMID 21471984
- [Background] Reich A, Orda A, Wisnicka B, Szepietowski JC. Plasma concentration of selected neuropeptides in patients suffering from psoriasis. Exp Dermatol. 2007 May;16(5):421-8. doi: 10.1111/j.1600-0625.2007.00544.x. PMID 17437485
- [Background] He Y, Ding G, Wang X, Zhu T, Fan S. Calcitonin gene-related peptide in Langerhans cells in psoriatic plaque lesions. Chin Med J (Engl). 2000 Aug;113(8):747-51. PMID 11776062
- [Background] Riol-Blanco L, Ordovas-Montanes J, Perro M, Naval E, Thiriot A, Alvarez D, Paust S, Wood JN, von Andrian UH. Nociceptive sensory neurons drive interleukin-23-mediated psoriasiform skin inflammation. Nature. 2014 Jun 5;510(7503):157-61. doi: 10.1038/nature13199. Epub 2014 Apr 23. PMID 24759321
- [Background] Kashem SW, Riedl MS, Yao C, Honda CN, Vulchanova L, Kaplan DH. Nociceptive Sensory Fibers Drive Interleukin-23 Production from CD301b+ Dermal Dendritic Cells and Drive Protective Cutaneous Immunity. Immunity. 2015 Sep 15;43(3):515-26. doi: 10.1016/j.immuni.2015.08.016. PMID 26377898
- [Background] Ding W, Stohl LL, Xu L, Zhou XK, Manni M, Wagner JA, Granstein RD. Calcitonin Gene-Related Peptide-Exposed Endothelial Cells Bias Antigen Presentation to CD4+ T Cells toward a Th17 Response. J Immunol. 2016 Mar 1;196(5):2181-94. doi: 10.4049/jimmunol.1500303. Epub 2016 Feb 1. PMID 26829986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the dermatology practices of the Weill Cornell Medical College Department of Dermatology and the practice of Neil Sadick, M.D., a voluntary faculty member of the department.
Pre-assignment Details: Ninety-six subjects were screened, 41 met criteria for entry. Five subjects withdrew or were withdrawn before being assigned to a group.
Period: Double-Blind Placebo Controlled Trial
Arm/Group | Rimegepant | Placebo | Rimegepant Extension-Previously Received Rimegepant-Open Label | Rimegepant Extension-Previously Received Placebo-Open Label
Started | 18 | 18 | 0 | 0
Completed | 17 (Number who completed Visit 9 (Week 16).) | 13 (Number who completed Visit 9 (Week 16).) | 0 | 0
Not Completed | 1 | 5 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Period: Extension Study
Arm/Group | Rimegepant | Placebo | Rimegepant Extension-Previously Received Rimegepant-Open Label | Rimegepant Extension-Previously Received Placebo-Open Label
Started | 0 | 0 | 12 | 6
Completed | 0 | 0 | 11 | 5
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rimegepant | Placebo | Rimegepant Extension-Previously Received Rimegepant-Open Label | Rimegepant Extension-Previously Received Placebo-Open Label | Total
Number analyzed (Participants) | 18 | 18 | 12 | 6 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number of subjects in each arm of the extension phase of our study are a subset of the subjects treated in the double blind, placebo controlled initial phase of the study.
  years
    Double-Blind Controlled Trial: number analyzed (Participants) | 18 | 18 | 0 | 0 | 36
    Double-Blind Controlled Trial | 47.72 (14.85) | 50.94 (14.09) |  |  | 49.29 (14.37)
    Open Label Extension: number analyzed (Participants) | 0 | 0 | 12 | 6 | 18
    Open Label Extension |  |  | 48.42 (15.29) | 46.33 (13.49) | 47.72 (14.34)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number of subjects in each arm of the extension phase of our study are a subset of the subjects treated in the double blind, placebo controlled initial phase of the study.
  Participants
    Double-Blind Controlled Trial: number analyzed (Participants) | 18 | 18 | 0 | 0 | 36
    Double-Blind Controlled Trial: Female | 6 | 6 |  |  | 12
    Double-Blind Controlled Trial: Male | 12 | 12 |  |  | 24
    Open Label Extension: number analyzed (Participants) | 0 | 0 | 12 | 6 | 18
    Open Label Extension: Female |  |  | 3 | 3 | 6
    Open Label Extension: Male |  |  | 9 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number of subjects in each arm of the extension phase of our study are a subset of the subjects treated in the double blind, placebo controlled initial phase of the study.
  Participants
    Double-Blind Controlled Trial: number analyzed (Participants) | 18 | 18 | 0 | 0 | 36
    Double-Blind Controlled Trial: Hispanic or Latino | 6 | 7 |  |  | 13
    Double-Blind Controlled Trial: Not Hispanic or Latino | 12 | 10 |  |  | 22
    Double-Blind Controlled Trial: Unknown or Not Reported | 0 | 1 |  |  | 1
    Open Label Extension: number analyzed (Participants) | 0 | 0 | 12 | 6 | 18
    Open Label Extension: Hispanic or Latino |  |  | 3 | 2 | 5
    Open Label Extension: Not Hispanic or Latino |  |  | 9 | 4 | 13
    Open Label Extension: Unknown or Not Reported |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number of subjects in each arm of the extension phase of our study are a subset of the subjects treated in the double blind, placebo controlled initial phase of the study.
  Participants
    Double-Blind Controlled Trial: number analyzed (Participants) | 18 | 18 | 0 | 0 | 36
    Double-Blind Controlled Trial: American Indian or Alaska Native | 0 | 0 |  |  | 0
    Double-Blind Controlled Trial: Asian | 1 | 2 |  |  | 3
    Double-Blind Controlled Trial: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Double-Blind Controlled Trial: Black or African American | 1 | 1 |  |  | 2
    Double-Blind Controlled Trial: White | 11 | 10 |  |  | 21
    Double-Blind Controlled Trial: More than one race | 0 | 0 |  |  | 0
    Double-Blind Controlled Trial: Unknown or Not Reported | 5 | 5 |  |  | 10
    Open Label Extension: number analyzed (Participants) | 0 | 0 | 12 | 6 | 18
    Open Label Extension: American Indian or Alaska Native |  |  | 0 | 0 | 0
    Open Label Extension: Asian |  |  | 1 | 1 | 2
    Open Label Extension: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0
    Open Label Extension: Black or African American |  |  | 0 | 1 | 1
    Open Label Extension: White |  |  | 7 | 4 | 11
    Open Label Extension: More than one race |  |  | 0 | 0 | 0
    Open Label Extension: Unknown or Not Reported |  |  | 4 | 0 | 4
Region of Enrollment [Number; unit: participants] — Population: The number of subjects in the double-blind, placebo controlled phase of the study is reported here.
  participants
    United States: number analyzed (Participants) | 18 | 18 | 0 | 0 | 36
    United States | 18 | 18 |  |  | 36
Region of Enrollment [Number; unit: participants] — Population: The number of subjects in the extension phase of the study is reported here.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 12 | 6 | 18
    United States |  |  | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Psoriasis as Measured by Percentage Change in the Psoriasis Area and Severity Index (PASI) Instrument
Description: Total score of Psoriasis Area and Severity Index ranges from 0 to 72. Change = (Week 16 score - Baseline score) for the placebo-controlled phase and (Week 15 score-Visit 12 score) for the extension phase. A low score means less severe disease while a high score reflects more severe disease. A score of 0 means no psoriasis. A PASI score of 5 to 10 is considered moderate disease and a score over 10 is considered severe. A score over 40 is rare.
  The primary outcome measure is the mean percent change in PASI score from baseline to week 16 in the placebo-controlled phase.
  For the extension phase, it is particularly interesting if a change is noted in the group that received placebo prior to the extension phase.
Time Frame: Baseline and Week 16 for placebo controlled trial. For Extension Phase, Visit 11/12 (Day 1) to Visit 15 (Week 12).
Population: The number of subjects in each arm of the extension phase of our study are a subset of the subjects treated in the double blind, placebo controlled initial phase of the study. Furthermore, one subject assigned to the placebo group was not included in the analysis due to having an adverse reaction (very severe insect bite reaction) prior to the first scheduled evaluation. Thus, the total number of analyzed subjects in the placebo-controlled phase was 35.
Measure: Mean (Standard Deviation); unit: Percent change in PASI score
Arm/Group | Rimegepant | Placebo | Rimegepant Extension-Previously Received Rimegepant-Open Label | Rimegepant Extension-Previously Received Placebo-Open Label
Number analyzed (Participants) | 18 | 17 | 12 | 6
Percent change in PASI score | 17.29 (34.43) | 27.06 (32.58) | 7.07 (31.68) | 20.02 (28.78)
Statistical Analysis 1: Comparison: Rimegepant vs Placebo; Test type: Superiority; p = 0.395, t-test, 2 sided — P value not adjusted for multiple comparisons,
Statistical Analysis 2: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label vs Rimegepant Extension-Previously Received Placebo-Open Label; Test type: Superiority; p = 0.410, t-test, 2 sided — P values not adjusted for multiple comparisons

2. Secondary Outcome: Number of Subjects Who Had a 50% or Greater Reduction in Psoriasis Area and Severity Index Instrument Score
Description: To record the number of subjects whose PASI Score Improves by at least 50% by week 16 (Week 16 average score - Baseline average score) for the placebo-controled phase and the change from Visit 12 (Day 1) to Visit 15 (Week 12) for the extension phase. PASI range is 0-72 although PASI must be at least 5 for entry into the study. A score of 0 means no psoriasis. A PASI score of 5 to 10 is considered moderate disease and a score over 10 is considered severe. A score over 40 is rare.
Time Frame: Baseline and Week 16 for placebo controlled trial. For Extension Phase, Visit 11/12 (Day 1) to Visit 15 (Week 12).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Rimegepant Extension-Previously Received Placebo-Open Label: Participants who previously received placebo receive a rimegepant 75 mg tablet orally every other day for an additional 12 weeks.
  Rimegepant: Active Agen
Arm/Group | Rimegepant | Placebo | Rimegepant Extension-Previously Received Rimegepant-Open Label | Rimegepant Extension-Previously Received Placebo-Open Label
Number analyzed (Participants) | 18 | 17 | 12 | 6
Participants | 3 | 4 | 1 | 0
Statistical Analysis 1: Comparison: Rimegepant vs Placebo; Test type: Superiority; p = 0.691, Fisher Exact
Statistical Analysis 2: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label vs Rimegepant Extension-Previously Received Placebo-Open Label; Test type: Superiority; p = 1, Fisher Exact — P values not adjusted for multiple comparisons

3. Secondary Outcome: Change in Severity of Psoriasis as Assessed by the Investigator's Global Assessment Instrument
Description: Score of the Investigator's Global Assessment instrument ranges from 0 to 5.
  Three parameters (erythema, induration and scaling, each is scored on a scale of 0 to 5. Erythema: 0 to 5 is the scale of intensity of erythema with 5 being the highest. Induration: 0 to 5 reflects the degree of elevation of the lesion with 5 being the most elevated. Scaling: 0 to 5 is the abundance of scale as well as the thickness and tenacious character of the scale with 5 being the most abundant, thick and tenacious scale) were each measured and averaged to obtain a score averaged to the nearest integer. The change from baseline to week 16 for each subject was calculated for the placebo-controlled phase and the change from Visit 12 to Visit 15 for the extension phase and the mean difference +/- standard deviation between groups was compared.
  For the extension phase, it is particularly interesting if a change is noted in the group that received placebo prior to the extension phase.
Time Frame: Baseline and Week 16 for placebo controlled trial. For Extension Phase, Visit 11/12 (Day 1) to Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rimegepant | Placebo | Rimegepant Extension-Previously Received Rimegepant-Open Label | Rimegepant Extension-Previously Received Placebo-Open Label
Number analyzed (Participants) | 18 | 17 | 12 | 6
score on a scale | 0.39 (0.98) | 0.47 (0.51) | 0.18 (0.40) | 0.5 (0.55)
Statistical Analysis 1: Comparison: Rimegepant vs Placebo; Test type: Superiority; p = 0.758, t-test, 2 sided; P value not adjusted for multiple comparisons,
Statistical Analysis 2: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label vs Rimegepant Extension-Previously Received Placebo-Open Label; Data represent change values; Test type: Superiority; p = 0.247, Fisher Exact — P values not adjusted for multiple comparisons

4. Secondary Outcome: Change in Dermatology Quality of Life Index
Description: Dermatology Quality of Life Index score ranges from 0-30. Average Change in Score of Each Group= (Week 16 average score - Baseline average score) for the placebo-controlled phase and (Visit 15 average score-Visit 12 average score) for the extension phase. 0 - 1 no effect at all on patient's life, 2 - 5 small effect on patient's life, 6 - 10 moderate effect on patient's life, 11 - 20 very large effect on patient's life, 21 - 30 extremely large effect on patient's life.
  For the extension phase, it is particularly interesting if a change is noted in the group that received placebo prior to the extension phase.
Time Frame: Baseline and Week 16 for placebo controlled trial. For Extension Phase, Visit 11/12 (Day 1) to Visit 15 (Week 12).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rimegepant | Placebo | Rimegepant Extension-Previously Received Rimegepant-Open Label | Rimegepant Extension-Previously Received Placebo-Open Label
Number analyzed (Participants) | 18 | 17 | 12 | 6
score on a scale | 2.22 (5.15) | 4.65 (8.4) | 1.45 (5.28) | 0.5 (2.07)
Statistical Analysis 1: Comparison: Rimegepant vs Placebo; Test type: Superiority; p = 0.316, t-test, 2 sided — P values were not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label vs Rimegepant Extension-Previously Received Placebo-Open Label; Data represent change values; Test type: Superiority; p = 0.605, t-test, 2 sided — P values not adjusted for multiple comparisons

5. Secondary Outcome: Change in Degree of Itching Assessed by the Visual Analogue Scale
Description: The Visual Analogue Scale ranges from 0 to 10. 0= no pruritus, < 3= mild pruritus, ≥ 3-<7= moderate pruritus, ≥ 7-<9 = severe pruritus, ≥ 9= very severe pruritus.
  We separately measured the reduction in average itch over the preceding 3 days and the reduction in maximum itch over the previous 7 days for each subject.
  For the extension phase, it is particularly interesting if a change is noted in the group that received placebo prior to the extension phase.
Time Frame: Baseline and Week 16 for placebo controlled trial. For Extension Phase, Visit 11/12 (Day 1) to Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rimegepant | Placebo | Rimegepant Extension-Previously Received Rimegepant-Open Label | Rimegepant Extension-Previously Received Placebo-Open Label
Number analyzed (Participants) | 18 | 17 | 12 | 6
score on a scale
  Mean reduction in average itch | 0.76 (2.64) | 2.05 (3.06) | 0.58 (2.01) | -0.07 (1.02)
  Mean reduction max itch | 0.93 (2.97) | 1.86 (2.81) | 0.43 (2.08) | -0.02 (1.09)
Statistical Analysis 1: Comparison: Rimegepant vs Placebo; Mean Reduction in Average Itch; Test type: Superiority; p = 0.192, t-test, 2 sided — P value not adjusted for multiple comparisons,
Statistical Analysis 2: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label vs Rimegepant Extension-Previously Received Placebo-Open Label; Mean Reduction in Average Itch. Data represent change values; Test type: Superiority; p = 0.392, t-test, 2 sided — P value not adjusted for multiple comparisons,
Statistical Analysis 3: Comparison: Rimegepant vs Placebo; Mean Reduction in Maximum Itch; Test type: Superiority; p = 0.347, t-test, 2 sided — P values not adjusted for multiple comparisons
Statistical Analysis 4: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label vs Rimegepant Extension-Previously Received Placebo-Open Label; Mean Reduction in Maximum Itch. Data represent change values; Test type: Superiority; p = 0.572, t-test, 2 sided — P value not adjusted for multiple comparisons,

6. Post Hoc Outcome: Median Change in the Psoriasis Area and Severity Index (PASI) Instrument Score From Visit 11/12 to Visit 15 in the Extension Phase - Previously Received Rimegepant Group
Description: Total score of Psoriasis Area and Severity Index ranges from 0 to 72. A low score means less severe disease while a high score reflects more severe disease. A score of 0 means no psoriasis. A PASI score of 5 to 10 is considered moderate disease and a score over 10 is considered severe. A score over 40 is rare. Change = (Week 15 score-Visit 12 score) for the extension phase was examined.
Time Frame: Visit 11/12 (Day 1) to Visit 15 (Week 12).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Rimegepant Extension-Previously Received Rimegepant-Open Label
Number analyzed (Participants) | 12
score on a scale | 0.9 [-3.0 to 5.2]
Statistical Analysis 1: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label; Test type: Other; p = 0.359, Wilcoxon (Mann-Whitney)

7. Post Hoc Outcome: Median Change in the Psoriasis Area and Severity Index (PASI) Instrument Score From Visit 11/12 to Visit 15 in the Extension Phase - Previously Received Placebo Group
Description: as for outcome 6
Time Frame: Visit 11/12 (Day 1) to Visit 15 (Week 12).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Rimegepant Extension-Previously Received Placebo-Open Label
Number analyzed (Participants) | 6
score on a scale | 1.35 [-1.69 to 5.8]
Statistical Analysis 1: Comparison: Rimegepant Extension-Previously Received Placebo-Open Label; Test type: Other; p = 0.141, Wilcoxon (Mann-Whitney)

8. Post Hoc Outcome: Median Change in the Dermatology Life Quality Index (DLQI) Instrument Score From Visit 11/12 to Visit 15 in the Extension Phase - Previously Received Rimegepant Group
Description: Dermatology Quality of Life Index score ranges from 0-30. . 0 - 1 no effect at all on patient's life, 2 - 5 small effect on patient's life, 6 - 10 moderate effect on patient's life, 11 - 20 very large effect on patient's life, 21 - 30 extremely large effect on patient's life. Change in Median Score of Each Group = (Visit 15 median score-Visit 11/12 median score) for the extension phase was examined
Time Frame: Visit 11/12 (Day 1) to Visit 15 (Week 12).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Rimegepant Extension-Previously Received Rimegepant-Open Label
Number analyzed (Participants) | 12
score on a scale | 0 [-6 to 14]
Statistical Analysis 1: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label; Test type: Other; p = 0.582, Wilcoxon (Mann-Whitney)

9. Post Hoc Outcome: Median Change in the Dermatology Life Quality Index (DLQI) Instrument Score From Visit 11/12 to Visit 15 in the Extension Phase - Previously Received Placebo Group
Description: as for outcome 8
Time Frame: Visit 11/12 (Day 1) to Visit 15 (Week 12).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Rimegepant Extension-Previously Received Placebo-Open Label
Number analyzed (Participants) | 6
score on a scale | 0.5 [-3 to 3]
Statistical Analysis 1: Comparison: Rimegepant Extension-Previously Received Placebo-Open Label; Test type: Other; p = 0.713, Wilcoxon (Mann-Whitney)

10. Post Hoc Outcome: Change in Severity of Psoriasis as Assessed by the Investigator's Global Assessment Instrument From Visit 11/12 to Visit 15 in the Extension Phase - Previously Received Rimegepant Group
Description: Score of the Investigator's Global Assessment instrument ranges from 0 to 5.
  Three parameters (erythema, induration and scaling, each is scored on a scale of 0 to 5. Erythema: 0 to 5 is the scale of intensity of erythema with 5 being the highest. Induration: 0 to 5 reflects the degree of elevation of the lesion with 5 being the most elevated. Scaling: 0 to 5 is the abundance of scale as well as the thickness and tenacious character of the scale with 5 being the most abundant, thick and tenacious scale) were each measured and averaged to obtain a score averaged to the nearest integer. The change from Visit 11/12 to Visit 15 for the extension phase was examined.
Time Frame: Visit 11/12 (Day 1) to Visit 15 (Week 12).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Rimegepant Extension-Previously Received Rimegepant-Open Label
Number analyzed (Participants) | 12
score on a scale | 0 [0 to 1]
Statistical Analysis 1: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label; Test type: Other; p = 0.346, Wilcoxon (Mann-Whitney)

11. Post Hoc Outcome: Change in Severity of Psoriasis as Assessed by the Investigator's Global Assessment Instrument From Visit 11/12 to Visit 15 in the Extension Phase - Previously Received Placebo Group
Description: as for outcome 10
Time Frame: Visit 11/12 (Day 1) to Visit 15 (Week 12).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Rimegepant Extension-Previously Received Placebo-Open Label
Number analyzed (Participants) | 6
score on a scale | 0.5 [0 to 1]
Statistical Analysis 1: Comparison: Rimegepant Extension-Previously Received Placebo-Open Label; Test type: Other; p = 0.149, Wilcoxon (Mann-Whitney)

12. Post Hoc Outcome: Change in Degree of Itching Assessed by the Visual Analogue Scale From Visit 11/12 to Visit 15 in the Extension Phase - Previously Received Rimegepant Group
Description: The Visual Analogue Scale ranges from 0 to 10. 0= no pruritus, < 3= mild pruritus, ≥ 3-<7= moderate pruritus, ≥ 7-<9 = severe pruritus, ≥ 9= very severe pruritus.
  We separately measured the reduction in average itch over the preceding 3 days and the reduction in maximum itch over the previous 7 days for each subject.
  Have examined the change in each score from visit 11/12 to visit 15 in the extension phase.
Time Frame: Visit 11/12 (Day 1) to Visit 15 (Week 12).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Rimegepant Extension-Previously Received Rimegepant-Open Label
Number analyzed (Participants) | 12
score on a scale
  Average Itch Preceding 3 Days | 0.6 [-3.6 to 4.5]
  Maximum Itch Within the Preceding 7 days | 0.4 [-4.5 to 3.5]
Statistical Analysis 1: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label; Analysis for Average Itch Over the Preceding 3 Days; Test type: Other; p = 0.221, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Rimegepant Extension-Previously Received Rimegepant-Open Label; Analysis is for the Maximum Itch of the Preceding 7 Days; Test type: Other; p = 0.286, Wilcoxon (Mann-Whitney)

13. Post Hoc Outcome: Change in Degree of Itching Assessed by the Visual Analogue Scale From Visit 11/12 to Visit 15 in the Extension Phase - Previously Received Placebo Group
Description: as for outcome 12
Time Frame: Visit 11/12 (Day 1) to Visit 15 (Week 12).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Rimegepant Extension-Previously Received Placebo-Open Label
Number analyzed (Participants) | 6
score on a scale
  Average Itch Preceding 3 Days | 0.05 [-1.7 to 1.4]
  Maximum Itch Within the Preceding 7 Days | 0 [-1.7 to 1.7]
Statistical Analysis 1: Comparison: Rimegepant Extension-Previously Received Placebo-Open Label; Analysis for Average Itch Over the Preceding 3 Days; Test type: Other; p = 1, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Rimegepant Extension-Previously Received Placebo-Open Label; Analysis is for the Maximum Itch of the Preceding 7 Days; Test type: Other; p = 1, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 20 weeks for the placebo-controlled phase for subjects that complete that phase and up to 34 weeks for subjects that enter the extension phase and completed it.
Description: One subject was withdrawn from the placebo group between the baseline visit and visit 1 due to an adverse reaction to bug bites. Therefore, the subject received IP and would be at risk for an AE but was not included in the analysis as we did not collect visit 1 data. Thus, for purposes of adverse events all 18 subjects assigned to the placebo group were included in the adverse events tables while only 17 subjects were included in the placebo-controlled phase in the outcome measures data tables.
Arm/Group | Rimegepant | Placebo | Rimegepant Extension-Previously Received Rimegepant-Open Label | Rimegepant Extension-Previously Received Placebo-Open Label
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 1/18 | 4/18 | 1/12 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rimegepant (N=18) | Placebo (N=18) | Rimegepant Extension-Previously Received Rimegepant-Open Label (N=12) | Rimegepant Extension-Previously Received Placebo-Open Label (N=6)
Acid Reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurry Vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Light Headedness Upon Standing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exaggerated Reaction to Insect Bites (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irregular Menses (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A relatively high number of subjects withdrew or were withdrawn. The were a relatively small number of subjects in the extension phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT04629950/Prot_SAP_000.pdf